CLINICAL TRIAL: NCT00005250
Title: Linkage Study of Long QT Syndrome In An Amish Kindred
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1132; R01HL041035 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-11

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Tachycardia, Ventricular; Ventricular Fibrillation; Long QT Syndrome
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Tachycardia, Ventricular; Ventricular Fibrillation; Long QT Syndrome

SUMMARY:
To screen by electrocardiography the entire population of 1,400 individuals in seven Amish Mennonite communities in order to perform genetic linkage studies of long QT syndrome (LQTS).

DETAILED DESCRIPTION:
BACKGROUND:

LQTS is a severe heart disorder leading to sudden death due to ventricular tachycardia or ventricular fibrillation. The syndrome segregated as a Mendelian recessive in the highly inbred population under study and resulted in the sudden death of several members of the population.

DESIGN NARRATIVE:

The entire population was screened to identify cases of LQTS. In addition, 29 obligate heterozygotes were studied by 24-hour Holter monitoring to determine whether these gene carriers had any subtle phenotypes. The data were subjected to complex segregation and linkage analysis to establish the mode of inheritance and penetrance of LQTS.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-01; Study Completion 1992-12 (Actual)